CLINICAL TRIAL: NCT05008159
Title: The Enhancing Physical and Community Mobility in Older Adults With Health Inequities Using Community Co-design of a Multifaceted Intervention Incorporating Physical Activity, Healthy Eating, Social Participation, and System Navigation (EMBOLDEN) Trial
Brief Title: A Community-based Program That Supports Physical Activity, Healthy Eating, Social Participation and System Navigation in Older Adults
Acronym: EMBOLDEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Labarge Centre for Mobility in Aging (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EMBOLDEN
Record Dates: First submitted 2021-07-29; First posted 2021-08-17 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Mobility Limitation; Health Related Quality of Life; Healthy Aging; Health Inequity
Keywords: Physical Mobility; Aging; Community-based intervention; Public and community engagement; Physical activity; Healthy eating; Social participation; System navigation; Life-space; Community mobility; Community integration
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Type II hybrid effectiveness-implementation RCT
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and interventionists are not blinded. All data collectors will be independent of the study and blinded to treatment allocation. Statisticians will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The EMBOLDEN program (Experimental): 3 month community-based mobility and healthy aging intervention
  Interventions: Behavioral: 3 month community-based mobility and health intervention
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: 3 month community-based mobility and health intervention — 12 weekly GROUP (10-15 adults per cohort) sessions + 3 INDIVIDUAL tailored system navigation sessions at beginning, midpoint, and end of program.
  The 3-month GROUP program will include the following fixed components:
  i) weekly interactive group-based health education sessions focused on:
  * increasing knowledge, skills, and behaviours related to physical activity, healthy eating, and available community supports for older adults;
  * socialization to foster peer and community connections, co-learning, and decrease social isolation
  * skill-building to support independence and quality of life; and
  ii) INDIVIDUAL tailored system navigation support
  Arms: The EMBOLDEN program

SUMMARY:
Physical mobility and social participation are needed to maintain independence and quality of life for adults over 55 years of age. Despite the known benefits of physical activity and dietary change programs for older adults, the best ways to deliver these interventions are not well understood. The goal of the EMBOLDEN study is to promote physical and community mobility in older adults who experience difficulties taking up community programs and reside in areas of high health inequity. Building on existing best practices, the investigators will implement and evaluate an innovative co-designed community-based program to promote physical activity, healthy eating, social participation, and system navigation. The potential for spreading this program throughout Hamilton and adapted to other Canadian communities will also be explored

DETAILED DESCRIPTION:
This is a randomized controlled trial employing a type II hybrid implementation-effectiveness design. This will enable the investigators to evaluate both clinical outcomes and important processes that impact the implementation of the co-designed intervention.

The intervention will consist of i) weekly interactive group-based health education sessions focused on: increasing knowledge, skills, and behaviours related to physical activity, healthy eating, and available community supports for older adults; this will include facilitated physical activity delivered by a certified exercise physiologist or certified personal trainer with experience and expertise working with older adults and interactive nutrition sessions; socialization to foster peer and community connections, co-learning, and decrease social isolation; and skill-building to support independence and quality of life; and ii) tailored system navigation support to increase access to and use of health and social services systems and address barriers or unmet needs

This trial has a pragmatic design in the following ways: i) recruiting a population with broad inclusion criteria, reflective of the general population of older adults; ii) conducting the study in existing community settings (when in-person delivery is feasible) and virtually, in partnership with organizations already delivering virtual supports due to the pandemic; iii) leveraging existing resources, staff, and service delivery organizations in the intervention arm that are available in usual care; iv) supporting flexibility delivery of the intervention (e.g., tailoring to participant group needs), as would be done through other community programs in usual care; v) flexibility in adherence to the intervention, in ways that are consistent with usual care; vi) selecting primary and secondary outcomes that are participant-relevant; and vii) using intention to treat analyses based on all available data.

The study will be delivered in community settings in urban neighbourhoods identified as areas of health inequities in the cities of Hamilton and Toronto, Ontario.

ELIGIBILITY:
Inclusion criteria:

• Community-dwelling older adults (55 years of age and older) living in a neighbourhood selected for the study.

Exclusion criteria:

* Unable to speak or understand English
* Unable to walk 10 meters without physical assistance from another person (assistive devices permitted)

As a pragmatic trial, we have chosen broad inclusion criteria to reflect the characteristics of individuals who may join a program such as this outside of a research study. Thus, we will not exclude individuals based on the presence of existing chronic disease, comorbidities, or other factors that may impact attendance.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Physical mobility | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in total weekly minutes spent in light, moderate-to-vigorous physical activity and sedentary activity as measured by an accelerometer worn over 7-day periods.

SECONDARY OUTCOMES:
Community mobility | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in community mobility as measured by GPS-derived quantity of out of home activities
Life Space mobility | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in life space mobility as measured by Life Space Index (LSI)which is a self-reported measure of community mobility with strong psychometric properties . Scores range from 0-120, where a score of 120 characterizes the highest possible level of life-space (i.e. going out of town without assistance). A change of 5 to 10 points on the LSI is considered clinically meaningful.
Physical activity | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in self-reported physical activity as measured by the Physical Activity Scale for the Elderly (PASE).
  PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.
Healthy eating and nutritional risk | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in healthy eating and nutritional risk as measured by Seniors in the community: risk evaluation for eating and nutrition, Version II (SCREEN-II). Scores range from 0 to 64. Lower scores on SCREEN II indicate increased risk for impaired nutritional states. Scores <50 indicate high nutrition risk.
Health-related quality of life | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in health-related quality of life as measured by the 12-Item Short Form Survey (SF-12). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Health-related quality of life | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in health-related quality of life as measured by the EQ-5D-5L. Scores range from -0.281 to 1, where values lower than 0 represent states considered to be worse than death. The instrument also includes a visual analogue scale (EQ-VAS) which provides a single global rating of self-perceived health and is scored on a 0 to 100 mm scale representing "the worst…" and "the best health you can imagine", respectively.
Loneliness | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in loneliness as measured by the 6-item De Jong Gierveld Loneliness scale. The total scale score is the sum of the item scores, ranging from 0 (not lonely) to 11 (extremely lonely). A score of 3 or higher is an indication of loneliness.
Depression | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in depression as measured by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
  Major depression is diagnosed if 5 or more of the 9 depressive symptom criteria have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. Other depression is diagnosed if 2, 3, or 4 depressive symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. One of the 9 symptom criteria ("thoughts that you would be better off dead or of hurting yourself in some way") counts if present at all, regardless of duration. As with the original PRIME-MD, before making a final diagnosis, the clinician is expected to rule out physical causes of depression, normal bereavement, and history of a manic episode.
Collective efficacy | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in the process of engaging and sustaining self-management support in everyday settings measured by the Collective Efficacy of Networks questionnaire (CENS). Scores can range from 12-60, with higher scores indicating higher self-management support.
Food security | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  2 questions validated from the US Department of Agriculture 18-item Household Food Security Survey (HFSS) that identifies risk for food insecurity if the participants answer that either or both of the following two statements is 'often true' or 'sometimes true' (vs. 'never true').
Community Belonging | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in sense of community belonging measured by social capital at the neighbourhood level. This is 1 question taken from the Canadian Community Health Survey: How would you describe your sense of belonging to your local community? Participants choose one of the following options: Very strong; Somewhat strong; Somewhat weak; Very weak.
Healthcare and social service utilization | Between baseline and 3-months. An additional comparison will be made at 6-months to examine whether potential changes are maintained in the post-intervention phase.
  Change in number of emergency room visits, number of hospitalizations, number of primary care and specialist visits.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ganann, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Community, Hamilton, Ontario(ON)
  - Downtown East Community, Toronto, Ontario(ON)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganann R, Phillips SM, Neil-Sztramko SE, Fisher K, Alvarez E, Kuspinar A, Newbold KB, Moore C, MacNeil M, Keller H, Teggart K, Thabane L, Agarwal G, Sherifali D, Adams J, Alshaikhahmed A. Study protocol for the randomized controlled trial of EMBOLDEN: a multifaceted intervention aimed at Enhancing physical and community MoBility in OLDEr adults with health inequities using commuNity co-design. Front Public Health. 2025 Apr 24;13:1555222. doi: 10.3389/fpubh.2025.1555222. eCollection 2025. PMID 40342494